CLINICAL TRIAL: NCT01609751
Title: Does a Daily Dose of the Probiotic Lactobacillus Casei Shirota Prevent Acute Episodes of Diverticulitis (LACTOPRoD) - a Pilot Study
Brief Title: Prevention of Diverticulitis by Taking a Daily Probiotic
Acronym: LACTOPRoD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPCRU2; Yakult UK (Other Grant/Funding Number: PO8959)
Record Dates: First submitted 2012-05-29; First posted 2012-06-01 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Acute Diverticulitis
Keywords: probiotic; lactobacillus; colonic diseases; dietary fibre
MeSH Terms: conditions — Colonic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Yakult 62 ml daily (Experimental)
  Interventions: Dietary Supplement: Yakult

INTERVENTIONS:
Dietary Supplement: Yakult — 62 ml dose daily for 365 days. There must be a cold chain from supplier (Yakult UK) via the primary care centre to the trial participants.
  Other Names: lactobacillus casei Shirota

SUMMARY:
There is evidence to show that daily probiotic Lactobacillus casei Shirota (LcS) in the form of Yakult fermented milk supports a healthy balanced population of "friendly" gut bacteria. This, coupled with evidence from four European trials showing probiotic benefit for recurrent diverticulitis and an understanding of how the disease develops, indicates that LcS may also be beneficial. The investigators plan to undertake a pilot study investigating whether consumption of once daily probiotic LcS as Yakult fermented milk would help either prevent attacks of diverticulitis completely or significantly reduce frequency of attacks. Subjects will be recruited from Surrey primary care units and will be closely monitored for 12 months whilst being supplied with a daily dose of for the full 12 months to see if this improves gut health.

DETAILED DESCRIPTION:
Because dietary fibre, obesity and diabetes are all confounding factors that influence the frequency and severity of attacks of diverticulitis, the research project will take account of this by:

1. Monitoring dietary fibre using a diet diary
2. Measurement of height and weight to determine BMI
3. Screening for undiagnosed diabetes and pre-diabetes

As well as keeping a diet diary, subjects will be asked to keep a general health diary, and to complete gut health questionnaires at start, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. A history of two episodes of UAD treated with antibiotics in the last five years.
2. Diverticulosis confirmed by colonoscopy, barium enema, USS, CT or MRI imaging or at surgery.
3. Agreement to consume one bottle of Yakult daily for 12 months
4. Availability of space in the domestic refrigerator for storage of Yakult units
5. Able to access depot (local primary care premises or chemist) to collect regular supplies of Yakult
6. Able to cope with keeping a diary etc.
7. Willing to take Yakult supplies and a cold bag on holiday to ensure as near as possible continuous daily doses (certainly never more than one week break as Lactobacilli casei will persist in the human gut for at least one week
8. Capable of giving informed consent
9. Aged ≥ 50 and ≤ 75 years at commencement of trial.

Exclusion Criteria:

1. Recent history of peptic ulcer
2. Chronic renal insufficiency
3. Ongoing or past major diverticulitis complications
4. Any serious debilitating illness (cancers, cardiovascular disease etc. but not DM)
5. Dementias or memory problems
6. Regular probiotic consumption over the past year.
7. Undergoing immunosuppressive therapy or treatment
8. Lactose intolerance or intolerance to dairy products
9. Immunosuppressed patients

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of episodes of acute diverticulitis | 12 months period of taking daily probiotic
  An episode of diverticulitis will be judged as having occured when there is left iliac pain and tenderness judged by the patient's genral practitioner to be due to acute diverticulitis and to be sufficiently severe as to require a course of antibiotics

SECONDARY OUTCOMES:
Gut symptoms assessed by a validated questionnaire at o months, 6 months and 12 months | 12 months
  The Bovenschen GIT symptom questionnaire (Bovenschen HJ, Janssen MJR, van Oijen MGH, Laheij RJF, van Rossum LGM, Jansen JBMJ (2006).Evaluation of Gastrolintestinal symptoms questionnaire. Digestive Diseases and Science;51:1509-1515.) will be used to assess this secondary endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Simon de Lusignan, MB ChB, Study Director — University of Surrey; John AA Nichols, MB ChB, Principal Investigator — University of Surrey; Michelle Gibbs, BSc PhD, Study Director — University of Surrey
Locations (1):
- Surrey Primary Care Trust practices, Guildford, Surrey, United Kingdom

REFERENCES:
- [Background] Narula N, Marshall JK. Role of probiotics in management of diverticular disease. J Gastroenterol Hepatol. 2010 Dec;25(12):1827-30. doi: 10.1111/j.1440-1746.2010.06444.x. PMID 21091992
- [Background] Annibale B, Maconi G, Lahner E, De Giorgi F, Cuomo R. Efficacy of Lactobacillus paracasei sub. paracasei F19 on abdominal symptoms in patients with symptomatic uncomplicated diverticular disease: a pilot study. Minerva Gastroenterol Dietol. 2011 Mar;57(1):13-22. PMID 21372765
- [Background] Bovenschen HJ, Janssen MJ, van Oijen MG, Laheij RJ, van Rossum LG, Jansen JB. Evaluation of a gastrointestinal symptoms questionnaire. Dig Dis Sci. 2006 Sep;51(9):1509-15. doi: 10.1007/s10620-006-9120-6. Epub 2006 Aug 22. PMID 16927133
- [Background] Hammerman C, Bin-Nun A, Kaplan M. Safety of probiotics: comparison of two popular strains. BMJ. 2006 Nov 11;333(7576):1006-8. doi: 10.1136/bmj.39010.630799.BE. No abstract available. PMID 17095783
- See also: Register using email address and search for "Find the science" then "Glossary" — http://hcp.yakult.co.uk